CLINICAL TRIAL: NCT07142603
Title: Comparative Meal Response to Plant vs. Animal Protein in Women With PCOS
Brief Title: Appetite Response to Meals With Different Protein Sources in Women With PCOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2507614944
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS; polycystic ovary syndrome; Protein; Women
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant protein challenge (Active Comparator): After an overnight fast, participants will be given a 350-400 kcal meal containing 30% energy from plant protein sources. Participants will be given 10 minutes to consume the meal and appetite and metabolic response will be measured for 240 following the meal.
  Interventions: Other: Metabolic response to protein source
- Animal Protein Challenge (Experimental): After an overnight fast, participants will be given a 350-400 kcal meal containing 30% energy from animal protein sources. Participants will be given 10 minutes to consume the meal and appetite and metabolic response will be measured for 240 following the meal.
  Interventions: Other: Metabolic response to protein source

INTERVENTIONS:
Other: Metabolic response to protein source — Participants will be given a 350-400 kcal meal challenge containing 30% energy from animal protein. They will be given 10 minutes to consume the meal and meal response will be measured 240 minutes following the meal.

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder characterized by insulin resistance, hyperandrogenism, and reproductive dysfunction. Dietary strategies that improve postprandial insulin and glucose responses are central to managing metabolic symptoms in PCOS.

Meals higher in protein can attenuate postprandial glycemia and enhance satiety, but the effects may vary by protein source. Animal sources of protein typically have higher essential amino acid content and insulinogenic potential, whereas plant proteins offer fiber and phytochemicals that may influence glycemic dynamics differently. Few studies have directly compared the acute metabolic effects of plant versus animal protein in women with PCOS. Given the distinct pathophysiology of PCOS, extrapolating findings from healthy populations may be misleading.

Understanding protein-specific effects on postprandial insulin, glucose, and appetite-regulating hormones in this group is essential for targeted nutrition guidance. Additionally, plant-based diets are increasingly promoted for cardiometabolic health, but their acute effects in insulin-resistant women remain underexplored. This study will assess whether plant and animal protein meals elicit differential postprandial responses in women with PCOS. Findings may inform dietary recommendations aimed at improving metabolic outcomes in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18-50 years
* Confirmed diagnosis of PCOS
* Body mass index (BMI) between 18.5 and 35 kg/m2
* Stable body weight for at least 3 months (+ 5 pounds)
* Willingness to consume both plant- and animal-based protein meals

Exclusion Criteria:

* Smoking or use of nicotine products
* Smoking or use of marijuana products
* Food allergies or dietary restrictions incompatible with test meals
* Diagnosed diabetes (type 1 or 2)
* Use of medications that interfere with study outcomes (e.g., metformin, GLP-1 agonists, etc.)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | Meal response over 240 minutes (0, 30, 60, 120, 180, and 240 minutes post meal challenge).
  Energy expenditure will be measured using indirect calorimetry.

SECONDARY OUTCOMES:
Appetite | Meal response over 240 minutes (0, 30, 60, 120, 180, and 240 minutes post meal challenge).
  Participants will be asked to rate their perceived hunger, fullness, and desire to eat with the use of a traditional 100 mm visual analog scales (VAS) with opposing anchors (e.g., "extremely hungry" or "not hungry at all"). The questions include "how hungry do you feel at this moment," "how full do you feel at this moment," "how strong is your desire to eat at this moment," and "how much food do you think you could eat at this moment." Participants will also be asked to evaluate the appearance ("how much do you like or dislike the appearance of the breakfast foods") and palatability ("how much do you like or dislike the smell and taste of the breakfast foods") of the breakfast with the use of a traditional 100 mm visual analog scale with opposing anchors "dislike extremely" or "like extremely." Appetite assessments were measured at 0, 15, 30, 60, 120, and 240 min after the meal.
Plasma amino acid response | Meal response over 240 minutes (0, 30, 60, 120, 180, and 240 minutes post meal challenge).
  Plasma amino acids will be measured using UPLC
Plasma biomarkers related to appetite | Meal response over 240 minutes (0, 30, 60, 120, 180, and 240 minutes post meal challenge).
  Appetite biomarkers including PYY (Peptide YY), CCK (cholecystokinin), BDNF (brain-derived neurotrophic factor), GLP-1 (glucagon-like petide-1), and ghrelin will be measured using commercially available kits. This measurements will be interpreted together to make a conclusion about a appetite regulation in response to protein source.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie I Baum, PhD, Principal Investigator — University of Arkansas, Fayetteville
Locations (1):
- Center for Human Nutrition, Fayetteville, Arkansas, United States